CLINICAL TRIAL: NCT07263451
Title: Safety and Feasibility of Irreversible Electroporation for Early-stage Breast Cancer: a Prospective, Open-Label, Single-Arm, Exploratory Study
Brief Title: Safety and Feasibility of IRE for Early-stage Breast Cancer: a Prospective, Open-Label, Single-Arm, Exploratory Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tian'an Jiang (Other)
Responsible Party: Sponsor-Investigator, Tian'an Jiang, Chief Physician, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IREBreast
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; IRE; Irreversible Electroporation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: To explore whether the irreversible electroporation can achieve the efficacy and feasibility of breast cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRE and Surgical Resection (Experimental): Qualified patients will receive IRE ablation, followed by standard surgical resection for breast cancer. The efficacy and feasibility of IRE will be evaluated through statistical analysis of the outcomes, which will be recorded in accordance with the primary and secondary efficacy endpoints.
  Interventions: Device: IRE by stunning pulse therapy device

INTERVENTIONS:
Device: IRE by stunning pulse therapy device — Qualified patients will receive IRE ablation, followed by standard surgical resection for breast cancer.During the process, patients will be followed up and evaluated

SUMMARY:
This is a prospective, open-label, single-arm, exploratory clinical trial conducted at our institution to investigate the use of Irreversible Electroporation (IRE) for the treatment of breast cancer.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, exploratory clinical trial conducted at our institution to investigate the use of Irreversible Electroporation (IRE) for the treatment of breast cancer. Qualified patients will receive IRE ablation, followed by standard surgical resection. The efficacy and feasibility of IRE will be evaluated through statistical analysis of the outcomes, which will be recorded in accordance with the primary and secondary efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18 years or older.
2. Medically fit for both surgery and general anesthesia, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. Treatment-naïve, primary, unifocal breast cancer with a maximum diameter of ≤ 2.0 cm as assessed by MRI.
4. Pathologically confirmed diagnosis of Invasive Ductal Carcinoma (IDC) within 3 months prior to enrollment.
5. Tumor that presents as a well-defined, localized mass and is clearly visualized on both breast ultrasound (for intraoperative guidance) and breast DCE-MRI (for baseline measurement and treatment planning).
6. The subject must be able to understand the purpose of the trial, voluntarily participate, and provide written informed consent.

Exclusion Criteria:

1. Known coagulopathy or bleeding diathesis (defined as a platelet count < 50×10⁹/L or an International Normalized Ratio (INR) > 1.5).
2. Presence of an implanted cardiac pacemaker, defibrillator, or any other active electronic medical device.
3. History of significant cardiac disease, including but not limited to: uncontrolled cardiac arrhythmias or congestive heart failure classified as New York Heart Association (NYHA) Class III or IV.
4. Patients who are pregnant, lactating, or planning a pregnancy during the study period.
5. Known severe allergy or anaphylactic reaction to MRI contrast agents.
6. Known high-risk genetic susceptibility to breast cancer (e.g., BRCA1/2 mutation carrier) associated with an increased risk of ipsilateral breast tumor recurrence following ablation.
7. Presence of distant metastases.
8. Any other medical or psychiatric condition that, in the investigator's judgment, would compromise the patient's safety or compliance with the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate | 1 month
  Pathologically confirmed absence of viable tumor cells in the resected tumor bed and margins of the post-IRE surgery specimen.
Technical success rate | 1 month
  The technical success rate of IRE ablation followed by surgery in treating breast cancer

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 month
  The incidence and severity of all adverse events (AE) and serious adverse events (SAE)
Pain scores | 1 month
  Pain scores of IRE ablation. The pain intensity was assessed using the 0-10 numerical rating scale (NRS), where 0 indicates no pain and 10 indicates the most severe pain.
Imaging analysis | 1 month
  the ablation lesion of the imaging results of the ablation lesion after IRE.

CONTACTS AND LOCATIONS:
Overall Officials: Tian'an Jiang, PhD, Study Chair — Zhejiang University; Peifen Fu, PhD, Study Chair — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zhang K, Teoh J, Laguna P, Dominguez-Escrig J, Barret E, Ramon-Borja JC, Muir G, Bohr J, de Reijke TM, Pelechano Gomez P, Ng CF, Sanchez-Salas R, de la Rosette J. Effect of Focal vs Extended Irreversible Electroporation for the Ablation of Localized Low- or Intermediate-Risk Prostate Cancer on Early Oncological Control: A Randomized Clinical Trial. JAMA Surg. 2023 Apr 1;158(4):343-349. doi: 10.1001/jamasurg.2022.7516. PMID 36723911
- [Background] Li S, Chen F, Shen L, Zeng Q, Wu P. Percutaneous irreversible electroporation for breast tissue and breast cancer: safety, feasibility, skin effects and radiologic-pathologic correlation in an animal study. J Transl Med. 2016 Aug 5;14(1):238. doi: 10.1186/s12967-016-0993-7. PMID 27495906
- [Background] Neal RE 2nd, Singh R, Hatcher HC, Kock ND, Torti SV, Davalos RV. Treatment of breast cancer through the application of irreversible electroporation using a novel minimally invasive single needle electrode. Breast Cancer Res Treat. 2010 Aug;123(1):295-301. doi: 10.1007/s10549-010-0803-5. Epub 2010 Feb 27. PMID 20191380
- [Background] Neal RE 2nd, Davalos RV. The feasibility of irreversible electroporation for the treatment of breast cancer and other heterogeneous systems. Ann Biomed Eng. 2009 Dec;37(12):2615-25. doi: 10.1007/s10439-009-9796-9. Epub 2009 Sep 15. PMID 19757056
- [Background] Collettini F, Enders J, Stephan C, Fischer T, Baur ADJ, Penzkofer T, Busch J, Hamm B, Gebauer B. Image-guided Irreversible Electroporation of Localized Prostate Cancer: Functional and Oncologic Outcomes. Radiology. 2019 Jul;292(1):250-257. doi: 10.1148/radiol.2019181987. Epub 2019 Jun 4. PMID 31161973
- [Background] Wang H, Xue W, Yan W, Yin L, Dong B, He B, Yu Y, Shi W, Zhou Z, Lin H, Zhou Y, Wang Y, Shi Z, Ren S, Gao X, Wang L, Xu C. Extended Focal Ablation of Localized Prostate Cancer With High-Frequency Irreversible Electroporation: A Nonrandomized Controlled Trial. JAMA Surg. 2022 Aug 1;157(8):693-700. doi: 10.1001/jamasurg.2022.2230. PMID 35793110
- [Background] Ruarus AH, Vroomen LGPH, Geboers B, van Veldhuisen E, Puijk RS, Nieuwenhuizen S, Besselink MG, Zonderhuis BM, Kazemier G, de Gruijl TD, van Lienden KP, de Vries JJJ, Scheffer HJ, Meijerink MR. Percutaneous Irreversible Electroporation in Locally Advanced and Recurrent Pancreatic Cancer (PANFIRE-2): A Multicenter, Prospective, Single-Arm, Phase II Study. Radiology. 2020 Jan;294(1):212-220. doi: 10.1148/radiol.2019191109. Epub 2019 Nov 5. PMID 31687922
- [Background] Al Efishat M, Wolfgang CL, Weiss MJ. Stage III pancreatic cancer and the role of irreversible electroporation. BMJ. 2015 Mar 18;350:h521. doi: 10.1136/bmj.h521. PMID 25787829
- [Background] Shankara Narayanan JS, Hayashi T, Erdem S, McArdle S, Tiriac H, Ray P, Pu M, Mikulski Z, Miller A, Messer K, Carson D, Schoenberger S, White RR. Treatment of pancreatic cancer with irreversible electroporation and intratumoral CD40 antibody stimulates systemic immune responses that inhibit liver metastasis in an orthotopic model. J Immunother Cancer. 2023 Jan;11(1):e006133. doi: 10.1136/jitc-2022-006133. PMID 36634919
- [Background] Timmer FEF, Geboers B, Ruarus AH, Vroomen LGPH, Schouten EAC, van der Lei S, Vos DJW, Dijkstra M, Schulz HH, Bakker J, van den Bemd BAT, van den Tol PM, Puijk RS, Lissenberg-Witte BI, de Gruijl TD, de Vries JJJ, Lagerwaard FJ, Scheffer HJ, Bruynzeel AME, Meijerink MR. MRI-guided stereotactic ablative body radiotherapy versus CT-guided percutaneous irreversible electroporation for locally advanced pancreatic cancer (CROSSFIRE): a single-centre, open-label, randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2024 May;9(5):448-459. doi: 10.1016/S2468-1253(24)00017-7. Epub 2024 Mar 19. PMID 38513683
- [Background] Distelmaier M, Barabasch A, Heil P, Kraemer NA, Isfort P, Keil S, Kuhl CK, Bruners P. Midterm Safety and Efficacy of Irreversible Electroporation of Malignant Liver Tumors Located Close to Major Portal or Hepatic Veins. Radiology. 2017 Dec;285(3):1023-1031. doi: 10.1148/radiol.2017161561. Epub 2017 Aug 11. PMID 28799842
- [Background] Sutter O, Calvo J, N'Kontchou G, Nault JC, Ourabia R, Nahon P, Ganne-Carrie N, Bourcier V, Zentar N, Bouhafs F, Sellier N, Diallo A, Seror O. Safety and Efficacy of Irreversible Electroporation for the Treatment of Hepatocellular Carcinoma Not Amenable to Thermal Ablation Techniques: A Retrospective Single-Center Case Series. Radiology. 2017 Sep;284(3):877-886. doi: 10.1148/radiol.2017161413. Epub 2017 Apr 28. PMID 28453431
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] Pan H, Yu M, Tang X, Mao X, Liu M, Zhang K, Qian C, Wang J, Xie H, Qiu W, Ding Q, Wang S, Zhou W. Preoperative single-dose camrelizumab and/or microwave ablation in women with early-stage breast cancer: A window-of-opportunity trial. Med. 2024 Apr 12;5(4):291-310.e5. doi: 10.1016/j.medj.2024.01.015. Epub 2024 Feb 27. PMID 38417440
- [Background] Geboers B, Scheffer HJ, Graybill PM, Ruarus AH, Nieuwenhuizen S, Puijk RS, van den Tol PM, Davalos RV, Rubinsky B, de Gruijl TD, Miklavcic D, Meijerink MR. High-Voltage Electrical Pulses in Oncology: Irreversible Electroporation, Electrochemotherapy, Gene Electrotransfer, Electrofusion, and Electroimmunotherapy. Radiology. 2020 May;295(2):254-272. doi: 10.1148/radiol.2020192190. Epub 2020 Mar 24. PMID 32208094
- [Background] Meijerink MR, Ruarus AH, Vroomen LGPH, Puijk RS, Geboers B, Nieuwenhuizen S, van den Bemd BAT, Nielsen K, de Vries JJJ, van Lienden KP, Lissenberg-Witte BI, van den Tol MP, Scheffer HJ. Irreversible Electroporation to Treat Unresectable Colorectal Liver Metastases (COLDFIRE-2): A Phase II, Two-Center, Single-Arm Clinical Trial. Radiology. 2021 May;299(2):470-480. doi: 10.1148/radiol.2021203089. Epub 2021 Mar 16. PMID 33724066
- [Background] Yu J, Han ZY, Li T, Feng WZ, Yu XL, Luo YC, Wu H, Jiang J, Wang JD, Liang P. Microwave Ablation Versus Nipple Sparing Mastectomy for Breast Cancer </=5 cm: A Pilot Cohort Study. Front Oncol. 2020 Oct 7;10:546883. doi: 10.3389/fonc.2020.546883. eCollection 2020. PMID 33117685
- [Background] Yang Q, Li H, Chen BH, He GZ, Wu XP, Wang LX, Wu H, Dou JP, Han ZY, Zhang J, Yu XL, Yu J, Liang P. Ultrasound-guided percutaneous microwave ablation for 755 benign breast lesions: a prospective multicenter study. Eur Radiol. 2020 Sep;30(9):5029-5038. doi: 10.1007/s00330-020-06868-9. Epub 2020 Apr 30. PMID 32356159
- [Background] Mauri G, Sconfienza LM, Pescatori LC, Fedeli MP, Ali M, Di Leo G, Sardanelli F. Technical success, technique efficacy and complications of minimally-invasive imaging-guided percutaneous ablation procedures of breast cancer: A systematic review and meta-analysis. Eur Radiol. 2017 Aug;27(8):3199-3210. doi: 10.1007/s00330-016-4668-9. Epub 2017 Jan 3. PMID 28050693
- [Background] Chu KF, Dupuy DE. Thermal ablation of tumours: biological mechanisms and advances in therapy. Nat Rev Cancer. 2014 Mar;14(3):199-208. doi: 10.1038/nrc3672. PMID 24561446
- [Background] Benson JR. Quality of life after breast-conserving surgery for women with non-low-risk ductal carcinoma in situ. Lancet Oncol. 2020 May;21(5):612-614. doi: 10.1016/S1470-2045(20)30135-2. Epub 2020 Mar 20. No abstract available. PMID 32203697
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636